CLINICAL TRIAL: NCT04780243
Title: Enhancing Postpartum Family Planning Utilization Through Integration With Expanded Program for Immunization in Sidama, South Ethiopia: A Quasi Experimental Study
Brief Title: Expanded Program for Immunization, a Missed Opportunity for Postpartum Family Planning Utilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hawassa University (Other)
Responsible Party: Principal Investigator, Abebaw Abeje Muluneh, Mr., Hawassa University
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: abe16muluneh
Record Dates: First submitted 2021-01-30; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention group (No Intervention): Pre-intervention group: women participated during the base line assessment will be labeled as Pre-intervention group
- postintervention group (Experimental): Postintervention group: women participated after the intervention was initiated will be labeled as postintervention group.
  Interventions: Other: counseling

INTERVENTIONS:
Other: counseling — Mothers presented to infant immunization units are going to be counseled for family planning services and if decide to take any method, they will be linked to family planning services
  Arms: postintervention group

SUMMARY:
This study is aimed to enhance postpartum family planning by integrating family planning information with infant immunization services, which is the most widely utilized health services globally.

DETAILED DESCRIPTION:
In this study, a before-and-after type of quasi-experimental study will be conducted in purposely selected health centers Sidama region, Ethiopia. base line assessment of postpartum contraceptive utilization rate will be done which will be followed by an intervention. The intervention consists of screening, counseling for family planning and referring mothers coming for infant immunization services to family planning units. All mothers coming for infant immunization service will be screened for and counseled for family planning and those who will be voluntary to take any method will be referred to family planning unit. All mothers who will not be voluntary will be re-counseled by the next visit.

Finally, the effect of this intervention on postpartum contraceptive utilization rate will be reassessed. The expected outcome will be to see an improved contraceptive uptake during the first year after delivery.

ELIGIBILITY:
Inclusion Criteria:

* all women visiting health facilities for infant immunization for at least two times will be included.

Exclusion Criteria:

* Women who are in difficulty of communicating during the study period will be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1474 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-03-17 (Estimated)

PRIMARY OUTCOMES:
After the initiation of the intervention, improved Contraceptive prevalence rate will be expected as an outcome | the outcome is measured two months after the initiation of the intervention
  After counseling of the postpartum mothers for family planning, their informed decision making capacity to use contraceptives will be increased.

CONTACTS AND LOCATIONS:
Overall Officials: Abebaw Muluneh, Principal Investigator — Hawassa University
Locations (1):
- Sidama regional health bureau, Awasa, Sidama Region, Ethiopia

IPD SHARING:
Plan to Share IPD: No